CLINICAL TRIAL: NCT06050070
Title: Targeting Large-scale Networks in Depression With Real-time fMRI Neurofeedback
Brief Title: Targeting Large-scale Networks in Depression With Real-time Functional Magnetic Resonance Imaging (fMRI) Neurofeedback
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Stephan F. Taylor, Professor of Psychiatry, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: HUM00228741 phase 3; 1R21MH134035-01 (NIH)
Record Dates: First submitted 2023-09-16; First posted 2023-09-22 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Major Depressive Disorder
Keywords: Functional MRI; Neurofeedback
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to sham or active feedback conditions, using block randomization stratified by gender, in a 50:50 allocation.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sham controlled feedback (Sham Comparator): Subjects will complete three visits with one or two fMRI sessions after initial assessment and training visit. The first session will be to introduce practice tasks using the mock scanner. In the second visit participants will have an fMRI. The study team will review the fMRI results to decide if participants will continue on the study (must exhibit a specific pattern of activation) and have the second fMRI at the third visit.
  Interventions: Other: FMRI with sham controlled feedback
- Real-time neurofeedback (Experimental): Subjects will complete three visits with one or two fMRI sessions after initial assessment and training visit. The first session will be to introduce practice tasks using the mock scanner. In the second visit participants will have an fMRI. The study team will review the fMRI results to decide if participants will continue on the study (must exhibit a specific pattern of activation) and have the second fMRI at the third visit.
  Interventions: Other: FMRI with real time feedback

INTERVENTIONS:
Other: FMRI with sham controlled feedback — During the second fMRI, the study will introduce the real time fMRI neurofeedback part of the study. This is where subjects will use the activity from the brain to control the size of the circular pattern viewed in the first two visits. This is real time fMRI because the pattern will change, in real time, based on what the fMRI scan measures in the brain. Participants will be encouraged to make the circular pattern grow in size, just by thinking about it.
  In order to see if the neurofeedback is really helping change the size of the circular pattern, the study team will have a control condition. In this controlled condition, subjects will see the circular pattern change, and the study team will ask participants to try and increase the size, except that the changing size will not actually be determined by your brain activity. This a called a sham condition because the feedback signal is not real.
  Arms: Sham controlled feedback
Other: FMRI with real time feedback — During the second fMRI, the study will introduce the real time fMRI neurofeedback part of the study. This is where subjects will use the activity from the brain to control the size of the circular pattern viewed in the first two visits. This is real time fMRI because the pattern will change, in real time, based on what the fMRI scan measures in the brain. Participants will be encouraged to make the circular pattern grow in size, just by thinking about it.
  Arms: Real-time neurofeedback

SUMMARY:
The purpose of this study is to develop a technique called real time fMRI neurofeedback.

This technique uses a regular MRI scanner, except that special software allows the researchers to measure activity in participants brain, using fMRI, and then give information, in the form of a feedback signal, which indicates brain activity in real time, while in the MRI scanner. The larger goal of this study is to develop ways to help people, including those with depression, better regulate brain activity. The researchers think that this may be helpful in managing psychiatric symptoms.

This study design has three phases, however, only two phases (phase 2 and 3) are considered to be a clinical trial. Phase 2 (part 2) was registered and is NCT05934604. This is the phase 3 (part 3) for this project and is funded by the National Institutes of Health.

DETAILED DESCRIPTION:
Part 3/Phase 3 study hypothesis are:

* Rest Focus Task (RFT) will activate brain networks at the individual subject level to provide a viable signal for Neurofeedback (NF)
* At the group level, RFT in the Active>Passive contrast will activate canonically defined salience network
* Neurofeedback-reinforced practice over the session will increase RFT activation over the course of the training session, comparing RFT activation, without NF, before and after NF runs.
* Valid Neurofeedback will increase RFT activation more compared to sham NF (assessed during the no-NF session).

ELIGIBILITY:
Inclusion Criteria:

* Meets The Diagnostic and Statistical Manual of Mental Disorders five (DSM5) criteria for Major Depressive Disorder, single or recurrent, active or in partial remission
* Patient Health Questionnaire (PHQ9) greater or equal (≥)6, and approximately (~) 50% with PHQ9≥10
* If participants are taking antidepressant medications, on stable dosage for 4 weeks
* No history of active substance use disorder in the past 6 months
* Absence of suicidal thoughts with plans or intentions, as assessed by Columbia Suicide Severity Rating Scale (C-SSRS)
* If a woman of child-bearing age, not pregnant or trying to become pregnant
* Ability to tolerate small, enclosed spaces without anxiety
* No metals, implants or metallic substances within or on the body that might cause adverse effects to the subject in a strong magnetic field, or interfere with image acquisition, e. g. aneurysm clips, retained particles (for example metal workers with exposures, protocol has more details), etc.
* Size compatible with scanner gantry (per protocol)
* Ability and willingness to give informed consent to participate.

Exclusion Criteria:

* Size not compatible with scanner
* Not meeting diagnostic criteria for bipolar disorder, schizophrenia, other psychosis, obsessive-compulsive disorder, active eating disorder or Post-traumatic stress disorder (PTSD)
* No history of serious neurological illness (including, but not limited to, seizures/epilepsy) or current medical condition that could compromise brain function, such as liver failure
* No history of closed head injury, e. g. loss of consciousness > ~5 min, hospitalization, neurological sequela

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-03-18 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Blood Oxygen Level Dependent (BOLD) signal change during the active > passive contrast during the localizer session | Approximately 40 minutes (during MRI)
  Using standard pre-processing pipelines, the general linear model, convolved with the hemodynamic response function, will be used to predict change in BOLD signal for the contrast of the active compared to the passive conditions. Z-transformed t-statistics will be corrected for multiple comparisons in the region of interest (salience network)
BOLD signal change during the active>passive contrast, comparing baseline with transfer runs (no NF in either), during the real time functional magnetic resonance imaging neurofeedback (rtfMRI-NF) session | Approximately 40 minutes (during MRI)
  Same processing as outcome measure 2, except the contrast of active>passive will itself be contrasted within the session (baseline compared to transfer run)

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Taylor, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No